CLINICAL TRIAL: NCT04410003
Title: Metabolic and Metagenomic Effects of Repopulation of the Intestinal Microbiome in Patients with Severe Unexplained Atherosclerosis
Brief Title: Metabolic and Metagenomic Effects of Intestinal Microbiome Repopulation in Unexplained Atherosclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: European Bioinformatics Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 115450
Record Dates: First submitted 2020-02-24; First posted 2020-06-01 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Atherosclerosis; Intestinal Microbiome
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients and persons involved in the followup and assessment of the participants will be blinded to the randomized assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Cellulose capsules, cloxacillin, electrolyte purgative (Peglyte)
  Interventions: Biological: Fecal microbial transplant
- Active (Active Comparator): Capsules of stool from Protected donors, cloxacillin, electrolyte purgative (Peglyte)
  Interventions: Biological: Fecal microbial transplant

INTERVENTIONS:
Biological: Fecal microbial transplant — Fecal microbial transplant

SUMMARY:
Patients with unexplained atherosclerosis (severe atherosclerosis not explained by traditional risk factors) will receive fecal microbial transplants (FMT) from patients with a Protected phenotype (patients who have high levels of risk factors but little or no carotid atherosclerosis). The objective is to determine what changes in the intestinal microbiome are associated with a decline in plasma levels of toxic metabolites of the itnestinal microbiome such as trimethylamine N-oxide (TMAO) and p-cresylsulfate. The intention is to develop an ecosystem therapeutic of cultured bacteria to treat atherosclerosis.

DETAILED DESCRIPTION:
100 patients with Unexplained Atherosclerosis, and 5 donors with the protected phenotype will be recruited; there will be extensive microbial, viral and parasitic screening of the donors. Recipients will be randomized to receive capsules of stool from the donors, or cellulose placebo. Recipients will take cloxacillin 500 mg 4 times daily for 5 days before the FMT, and will undergo purging with an electrolyte solution, (PegLyte) the day before the FMT. Metagenomic analysis of the recipient stool will be performed before FMT, 6 weeks later and after 12 months.Plasma levels of toxic intestinal metabolites will be measured before FMT, at 6 weeks and 12 months after FMT; the levels to be measured will be TMAO, P-cresylsulfate, Hippuric acid. Indoxyl sulfate, P-cresyl glucuronide. Phenyl acetyl glutamine, and Phenyl sulfate.

The investigators will analyze the metagenomic changes in the intestinal microbiome of recipients that are associated with decline in the plasma levels of the metabolic products of the intestinal microbiome to identify candidate bacteria for an "ecosystem therapeutic for atherosclerosis. Based on previous experience of designing such a therapeutic for clostridium difficile, it is anticipated that ~ 40 bacterial species would be needed.

ELIGIBILITY:
Inclusion Criteria:

* Severe atherosclerosis, with total plaque area in the top quartile (>119 mm2), not explained by traditional risk factors in linear regression (residual score >= 2)

Exclusion Criteria:

* Excluded will be patients unwilling/unable to provide informed consent, unwilling to ingest the stool capsules at baseline, patients with moderate to severe renal failure (eGFR<50), immunosuppressed patients, and patients with cancer, unstable angina, planned carotid revascularization or other conditions that might be expected to reduce their survival to < 1 year (including age >80).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma levels of metabolites of the intestinal microbiome | 6 weeks and 12 months
  The primary outcome is changes in plasma levels of trimethylamine N-oxide and p-cresylsulfate
Metagenomic changes of the intestinal microbiome | 6 weeks and 12 months
  Metagenomic changes in the stool of transplant recipients will be analyzed to determine what changes in the intestinal bacteria are associated with changes in the plasma levels of the intestinal metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: J. David Spence, M.D., Principal Investigator — Western University, Canada; Chrysi Bogiatzi, M.D., Study Director — Division of Neurology, Western University
Locations (1):
- Stroke Prevention & Atherosclerosis Research Centre, Robarts Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data might be made available with approval of the ethics committee

REFERENCES:
- [Background] Bogiatzi C, Gloor G, Allen-Vercoe E, Reid G, Wong RG, Urquhart BL, Dinculescu V, Ruetz KN, Velenosi TJ, Pignanelli M, Spence JD. Metabolic products of the intestinal microbiome and extremes of atherosclerosis. Atherosclerosis. 2018 Jun;273:91-97. doi: 10.1016/j.atherosclerosis.2018.04.015. Epub 2018 Apr 17. PMID 29702430